CLINICAL TRIAL: NCT02046447
Title: Neuroimaging of Dystonia: The Bachmann-Strauss Dystonia and Parkinson Disease Center of Excellence at the University of Florida
Brief Title: Neuroimaging of Dystonia
Acronym: NID
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Bachmann Strauss Dystonia & Parkinson Foundation, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 354-2013
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Primary Cervical Dystonia; DYT 1 Dystonia
Keywords: dystonia; cervical dystonia; DYT1; DYT 1; DYT-1; Dystonia 1; fMRI; healthy; trihexyphenidyl; Artane; Apo-Trihex; Parkin; Pacitane; Benzhexol; Trihex
MeSH Terms: conditions — Cervical Dystonia, Primary; Dystonia; Torticollis; Dystonia musculorum deformans type 1; Dystonia Musculorum Deformans | interventions — Trihexyphenidyl; Ubiquitin-Protein Ligases; trihex

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Primary Cervical Dystonia (Trihexyphenidyl): These subjects will receive the following: 1) data about clinical movement disorder history, age, gender, height, weight, and other medical conditions; 2) clinical neurological examination; 3) tests assessing cognitive abilities including: the Montreal Cognitive Assessment, Stroop, Digit Span, and Brief Test of Attention (BTA); 4) measures of anxiety and depression: the Beck Depression Index (BDI II). Only participants aged 18+ will be given the BDI; and 5) Functional magnetic resonance imaging (fMRI) and structural MRI will be performed.
  After the above baseline testing these subjects will receive a dose of trihexyphenidyl 2 mg an hour prior to the second functional fMRI scan. The subjects will be done with the study after the second MRI scan has been completed.
  Interventions: Drug: Primary Cervical Dystonia (Trihexyphenidyl)
- DYT 1 Dystonia (Healthy Control): These subjects will receive the following: 1) data about clinical movement disorder history, age, gender, height, weight, and other medical conditions; 2) clinical neurological examination; 3) tests assessing cognitive abilities including: the Montreal Cognitive Assessment, Stroop, Digit Span, and Brief Test of Attention (BTA); 4) measures of anxiety and depression: the Beck Depression Index (BDI II). Only participants aged 18+ will be given the BDI; and 5) Functional magnetic resonance imaging (fMRI) and structural MRI will be performed.
  Interventions: Other: DYT 1 Dystonia (Healthy Control)
- Primary Cervical Dystonia (Healthy Control): These subjects will receive the following: 1) data about clinical movement disorder history, age, gender, height, weight, and other medical conditions; 2) clinical neurological examination; 3) tests assessing cognitive abilities including: the Montreal Cognitive Assessment, Stroop, Digit Span, and Brief Test of Attention (BTA); 4) measures of anxiety and depression: the Beck Depression Index (BDI II). Only participants aged 18+ will be given the BDI; and 5) Functional magnetic resonance imaging (fMRI) and structural MRI will be performed.
  Interventions: Other: Controls Primary Cervical Dystonia (Trihexyphenidyl)
- DYT 1 Dystonia: These subjects will receive the following: 1) data about clinical movement disorder history, age, gender, height, weight, and other medical conditions; 2) clinical neurological examination; 3) tests assessing cognitive abilities including: the Montreal Cognitive Assessment, Stroop, Digit Span, and Brief Test of Attention (BTA); 4) measures of anxiety and depression: the Beck Depression Index (BDI II). Only participants aged 18+ will be given the BDI; 5) Functional magnetic resonance imaging (fMRI) and structural MRI will be performed; and 6) Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) to assess dystonia severity.
  Interventions: Other: DYT 1 Dystonia

INTERVENTIONS:
Drug: Primary Cervical Dystonia (Trihexyphenidyl) — After the baseline testing these subjects will receive a dose of trihexyphenidyl 2 mg an hour prior to the second functional magnetic resonance imaging (fMRI) scan. This is to test the change in cerebral blood flow based on blood-oxygen-level dependent (BOLD) contrast during a precision gripping task after administration of trihexyphenidyl compared to change in BOLD contrast during a precision gripping task. The subjects will be done with the study after the second MRI scan has been completed.
  Other Names: Artane; Apo-Trihex; Parkin; Pacitane; Benzhexol; Trihex; Trihexphenidyl
  Groups: Primary Cervical Dystonia (Trihexyphenidyl)
Other: Controls Primary Cervical Dystonia (Trihexyphenidyl) — These subjects will receive the following: 1) data about clinical movement disorder history, age, gender, height, weight, and other medical conditions; 2) clinical neurological examination; 3) tests assessing cognitive abilities including: the Montreal Cognitive Assessment, Stroop, Digit Span, and Brief Test of Attention (BTA); 4) measures of anxiety and depression: the Beck Depression Index (BDI II). Only participants aged 18+ will be given the BDI; and 5) Functional magnetic resonance imaging (fMRI) and structural MRI will be performed.
  Groups: Primary Cervical Dystonia (Healthy Control)
Other: DYT 1 Dystonia (Healthy Control) — These subjects will receive the following: 1) data about clinical movement disorder history, age, gender, height, weight, and other medical conditions; 2) clinical neurological examination; 3) tests assessing cognitive abilities including: the Montreal Cognitive Assessment, Stroop, Digit Span, and Brief Test of Attention (BTA); 4) measures of anxiety and depression: the Beck Depression Index (BDI II). Only participants aged 18+ will be given the BDI; and 5) Functional magnetic resonance imaging (fMRI) and structural MRI will be performed.
  Groups: DYT 1 Dystonia (Healthy Control)
Other: DYT 1 Dystonia — These subjects will receive the following: 1) data about clinical movement disorder history, age, gender, height, weight, and other medical conditions; 2) clinical neurological examination; 3) tests assessing cognitive abilities including: the Montreal Cognitive Assessment, Stroop, Digit Span, and Brief Test of Attention (BTA); 4) measures of anxiety and depression: the Beck Depression Index (BDI II). Only participants aged 18+ will be given the BDI; and 5) Functional magnetic resonance imaging (fMRI) and structural MRI will be performed.
  Groups: DYT 1 Dystonia

SUMMARY:
The main purpose of this study is to investigate primary cervical dystonia as compared to healthy control subjects and DYT 1 dystonia as compared to healthy control subjects by examining cognitive measures, physical measures, and structural and functional magnetic resonance imaging (MRI).

The secondary aim of this study is to investigate a specific drug therapy for primary cervical dystonia to develop a functional MRI (fMRI) research paradigm. The drug, trihexyphenidyl, is FDA approved to treat Parkinson's Disease and is commonly prescribed by physicians as a treatment for symptoms of primary cervical dystonia.

DETAILED DESCRIPTION:
To participate in this study, you will be asked to come to the University of Florida for one testing day. For your convenience, arrangements will be made by the study coordinator.

If you have a movement disorder, you will be tested in an "off" medication condition. We do not expect concerns or unwanted consequences arising from discontinuing medications for this duration.

We will review the informed consent and you will have the opportunity to ask questions before signing the informed consent. During the experiment, you may be asked to complete the following: (1) questionnaires about quality of life and depression; (2) tests to measure your strength and motor function; (3) tests to measure your cognition; (4) functional and structural MRI scan of your brain while performing a precision gripping task; (5) intravenous blood draw; (6) urine pregnancy test (if applicable); (7) trial of anticholinergic therapy drug trihexyphenidyl (if applicable - cervical dystonia only).

Participants with DYT 1 dystonia and healthy controls are not eligible to receive the trial drug. All women of childbearing potential will be given a urine pregnancy test. The questionnaire about depression will not be given to subjects under the age of 18.

If you have any metal in your eye or eyes, the researchers may require additional screening to ensure that it is safe for you to enter the MRI environment. If additional screening is determined to be necessary, you will be referred to Radiology at Shands UF for an orbitofrontal x-ray.

Blood will be collected for all subjects, including healthy control subjects. The blood may be analyzed, at the University of Florida, to assess potential biomarkers for cervical dystonia and DYT 1 dystonia. Biomarker testing is another way to say genetic testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary cervical dystonia and between the ages of 18-70, OR
* Diagnosis of DYT 1 dystonia and between the ages of 7-50, OR
* Healthy control and between the ages of 7-70

Exclusion Criteria:

* Neurological impairment from: seizure disorders, stroke, hypertension, heart disease, diabetes, traumatic brain injury (TBI), drug abuse, nerve disorders, dementia, Parkinson's Disease, dementia
* Not a candidate for magnetic resonance imaging (MRI)
* Deep brain stimulation (DBS) surgery
* Any implanted electrical device
* Pregnant or planning pregnancy
* Breastfeeding
* Claustrophobia

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Qualifying candidates with a diagnosis of DYT 1 dystonia will be identified and invited to participate utilizing an IRB approved database and neurologists review.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in cerebral blood flow based on blood-oxygen-level dependent (BOLD) contrast during a precision gripping task | 1 hour
  Participants will use their hand to squeeze an MRI compatible grip force transducer in the MRI unit. While producing force, the participants will observe the amount of force generated by viewing a visual feedback display.
Change in cerebral blood flow based on blood-oxygen-level dependent (BOLD) contrast during a precision gripping task after administration of trihexyphenidyl compared to change in BOLD contrast during a precision gripping task | 2 hours
  Subjects with primary cervical dystonia will repeat the primary outcome measure "Change in cerebral blood flow based on blood-oxygen-level dependent (BOLD) contrast during a precision gripping task" one hour after administration of 2mg trihexyphenidyl tablet.

CONTACTS AND LOCATIONS:
Overall Officials: David Vaillancourt, PhD, Principal Investigator — University of Florida; Michael Okun, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- See also: Tyler's Hope for a Dystonia Cure — http://www.tylershope.org/
- See also: UF Center for Movement Disorders & Neurorestoration — http://movementdisorders.ufhealth.org/